CLINICAL TRIAL: NCT06107751
Title: Comparison of Ramped and Sniffing Positions in Video-laryngoscopy-guided Tracheal Intubation for Elective Cesarean Section: a Prospective Randomized Study.
Brief Title: Ramped and Sniffing Position for Cesarean Section Intubation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, muhammet korkusuz, Principal Investigator, MD, Karaman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-2023/14
Record Dates: First submitted 2023-10-20; First posted 2023-10-30 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Intubation; Difficult or Failed
Keywords: Cesarean section; Intubation; Videolaryngoscopy

STUDY DESIGN:
Intervention Model Description: There are two group;
  1. Experimental Group: Group R; Ramped Group; Pillows will be placed under the patient's upper body and head, with the external auditory canal and sternal notch horizontal.
  2. Sham Comparator: Group S; Sniffing Group; A 7 cm high pillow will be placed under the occiput while the patient is in the supine position.
Who Masked: Participant, Care Provider
Masking Description: Due to the nature of the study, patients and care providers will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramped position group (Active Comparator): This position will be achieved by elevation of the shoulders and the head elevation till achieving alignment of sternal notch and external auditory meatus
  Interventions: Other: Ramped position group
- Sniffing position group (Sham Comparator): This position will be achieved by placing a 7 cm pillow under the occiput.
  Interventions: Other: Sniffing position group

INTERVENTIONS:
Other: Ramped position group — This position will be achieved by elevation of the shoulders and the head elevation till achieving alignment of sternal notch and external auditory meatus
  Other Names: Ramped position
  Arms: Ramped position group
Other: Sniffing position group — This position will be achieved by placing a 7 cm pillow under the occiput.
  Other Names: Sniffing group
  Arms: Sniffing position group

SUMMARY:
This study will include pregnants who preferred to undergo general anesthesia for elective cesarean section. Ramped and sniffing positions of pregnant women during ventilation and intubation will be compared. The aim of this study is to investigate which position provides easier and faster intubation in pregnant women for cesarean section.

DETAILED DESCRIPTION:
Estimates of the frequency of difficult and failed intubation in the obstetric population vary within a wide range of percentiles. Several times higher than those reported for the general surgery population. Functional Residual Capacity decreases by 10% - 25% in Pregnant women. Pregnant women are more susceptible to hypoxia as a result of this decline, which also encourages intubation to occur more rapidly. Intubation success and shortening of intubation time have improved positively with videolaryngoscopes. On the other hand, the position of the patient during intubation contributes to the speed and success of intubation. It has been shown that intubation is faster and first-pass success is higher in the ramped position in morbidly obese patients.This study will compare the effectiveness of ramp and sniffing positions on intubation time and success in obese patients and pregnant women with similar physical changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status classification of II-III, who are planned for elective cesarean section, who are between the ages of 18 and 40, and who prefer general anesthesia will be included.

Exclusion Criteria:

* Patients who refuse to participate in the study, have orientation and cooperation disorders, have undergone head and neck surgery, have a history of difficult intubation, have a cervical spine defect, and have a risk of pulmonary aspiration will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since intubation time for cesarean section will be evaluated, only female patients will be studied.
Enrollment: 60 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
1. Total intubation time | 5 minutes after induction of general anesthesia
  Total intubation time will be calculated by adding up the laryngoscopy time and tube insertion time.

SECONDARY OUTCOMES:
Incidence of difficult intubation | 5 minutes after induction of general anesthesia
  The Intubation Difficulty Scale (IDS) will be used to define the intubation difficulty. Intubation is considered easy if IDS=0, slight difficulty if 0 < IDS < 5, Moderate to Major Difficulty if 5 < IDS, impossible if IDS = ∞.
Incidence of difficult mask ventilation | 5 minutes after induction of general anesthesia
  The Warters Scale will be used to define the mask ventilation difficulty. Difficult mask ventilation is defined as a score ≥ 4 on the Warters scale
Laryngoscopy time | 5 minutes after induction of general anesthesia
  The timing measurements will begin when the videolaryngoscope blade first passes between the teeth and will end when the best glottic view is obtained on the videolaryngoscopy monitor.
Tube insertion time | 5 minutes after induction of general anesthesia
  The timing measurements will begin when the endotracheal tube first passes between the teeth and ended when the tube passes through the glottis.
Complications related to intubation | postoperative 4th hour
  A postoperative follow-up assessment will be performed approximately 4 hr after surgery by a co-investigator blinded to the intubation position to evaluate the presence and severity of sore throat, any changes in voice, trauma to the lip, tongue, palate, or teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, MD, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)